CLINICAL TRIAL: NCT03820661
Title: Advancing The Local Staging Of Pancreatic Ductal Adenocarcinoma Through High-Resolution Ultrasound: A Pilot Study
Brief Title: High Resolution Ultrasound in Pancreatic Ductal Adenocarcinoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18-5982
Record Dates: First submitted 2019-01-11; First posted 2019-01-29 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Resolution Ultasound (Other): Diagnostic high resolution ultrasound pre-operatively and intraoperatively
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — High resolution ultrasound pre-operatively and intra-operatively

SUMMARY:
Pancreatic cancer patients at UHN who have had a CT at UHN and have surgery planned will undergo a high resolution ultrasound pre-operatively and intra-operatively. This study is being done to see if using high resolution ultrasound before and during surgery will help the doctors accurately diagnose pancreatic ductal adenocarcinoma and identify if the disease has spread to other areas of the body.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females > 18 y
2. PDAC diagnosed by typical imaging findings or pathology
3. Scheduled for surgical resection
4. Contrast enhanced CT scan performed locally at UHN

Exclusion Criteria:

1) Inability or unwillingness to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
High-resolution U/S will be used to measure vascular invasion and regional lymph node metastases in PDAC | within 2 weeks of surgery
  The U/S results will be compared to pre-operative CT scan to help determine the diagnostic effectiveness of High Resolution US

CONTACTS AND LOCATIONS:
Overall Officials: Korosh Khalili, MD, Principal Investigator — UHN
Locations (1):
- University Health Network, Toronto, Ontario, Canada